CLINICAL TRIAL: NCT03913650
Title: Preoperative Peripheral Nerve Blocks Attenuate Intraoperative Surgical Stress and Postoperative Pain in Patients Undergoing Orthopedic Surgery
Brief Title: The Influence of Peripheral Nerve Blocks in Patients Undergoing Limb Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Municipal Hsiaokang Hospital (Other Government)
Responsible Party: Principal Investigator, I-Cheng Lu, Visiting staff, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUH-IRB-F(I)-20170007
Record Dates: First submitted 2017-09-17; First posted 2019-04-12 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative; Change; Circulatory; Surgical Injury
Keywords: peripheral nerve block; IL-6; post-operative pain; limb surgery
MeSH Terms: conditions — Pain, Postoperative; Intraoperative Complications | interventions — Bupivacaine; Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nerve block(+) (Active Comparator): patient accept nerve block for post-op pain control
  Interventions: Procedure: 0.25% bupivacaine
- Morphine (Sham Comparator): patient received morphine for post-op pain control
  Interventions: Procedure: 0.25% bupivacaine

INTERVENTIONS:
Procedure: 0.25% bupivacaine — nerve block procedure will be decided by patients' will for post-op pain
  Other Names: nerve block with 0.25% bupivacaine

SUMMARY:
To investigate pre-op peripheral nerve block in reducing peri-op IL-6 level and post-op pain

DETAILED DESCRIPTION:
In orthopedic surgery, peripheral nerve block can be used as an anesthesia adjuvant prior to surgery. In this study, we hypothesized that peripheral nerve blocks may alleviate inflammatory response and reduce the analgesics requirement. Sixty patients undergoing limb orthopedic surgery will be enrolled. Peripheral nerve block was injected with 0.25% bupivacaine under ultrasound guidance. 30 patients (Study group) underwent surgery with nerve blocks and another 30 patients (Control group) underwent surgery with morphine. The anesthetic protocol was standardized for both groups by experienced anesthesiologists. Surgical stress was assessed by blood pressure fluctuation and proinflammatory cytokine. Pain intensity was measured by numeric rating scale (NRS) score for 24 hours

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of limb fracture
* must receiving orthopedic surgery

Exclusion Criteria:

* With the comorbidity of chronic heart, lung, liver and renal disease, Chronic alcoholism, Allergy to bupivacaine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
peak pain intensity in the postoperative care unit | 2 hours
  pain score evaluated by pain score

SECONDARY OUTCOMES:
change of perioperative IL-6 level | up to 6 hours
  blood samples assessed by ELISA

OTHER OUTCOMES:
changes of perioperative hemodynamic parameter | up to 3 hours
  heart rate
changes of perioperative hemodynamic parameter | up to 3 hours
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: I-Cheng Lu, MD, PHD, Study Chair — Kaohsiung Medical University
Locations (2):
- Taiwan (2):
  - I-Cheng Lu, Kaohsiung City
  - Kaohsiung Municipal Siaogang Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: Undecided